CLINICAL TRIAL: NCT03459547
Title: Features of Peri-implant Soft Tissue Early Healing Around Different Abutment Materials
Brief Title: Soft Peri-implant Tissue Around Different Abutment Materials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Max-Planck Institute of Molecular Cell Biology and Genetics (Other)
Responsible Party: Principal Investigator, Andrea Pilloni MD DDS MS, MD DDS MS, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000102
Record Dates: First submitted 2018-02-07; First posted 2018-03-09 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Dental Implant Failure Nos; Wound Heal
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: Patients of more than 18 years old without systemic disease/ disorders, smokers of less 5 cigarettes per day, periodontally healthy or treated with full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) ≤ 15% at baseline with edentulous space needing an all on four or all on six treatment with overdenture width of the keratinized gingiva ≥ 2 at the level of the crest
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- dental implant + PEEK (test) (Experimental): Dental implant insertion, material polyetheretherketone
  Interventions: Device: dental implant
- dental implant + Ti-5 (control) (Active Comparator): Dental implant insertion, material titanium group 5
  Interventions: Device: dental implant
- dental implant + zirconia (control) (Active Comparator): dental implant insertion, material zirconia
  Interventions: Device: dental implant
- dental implant + Ti-4 (control) (Active Comparator): dental implant insertion, material titanium group 4
  Interventions: Device: dental implant

INTERVENTIONS:
Device: dental implant — Local anesthesia, flap preparation, dental implant insertion, flap suture, healing abutment insertion. Peri-implant soft tissue samples taken prior to implant placement and 24 hours after.
  Other Names: PEEK; Ti-4; Ti-5; zirconia

SUMMARY:
Soft tissue attachment to the implant surface serves as a biological seal preventing the development of inflammatory periimplant diseases (i.e. peri-implant mucositis and peri-implantitis).It occurs in the presence of a biomaterial during healing of the surgical wound that might be influence by this foreign body. Myofibroblasts represent key players in the physiological reconstruction of connective tissue after injury.

This work will focus on the role of myofibroblasts during the early phases of the healing process in peri-implant tissues around four different abutment materials.

DETAILED DESCRIPTION:
Dental implants are anchored in jawbone through a direct bonding between bone and the implant. Success and survival of an implant do, however, not depend solely on osseointegration. A soft tissue, which surrounds the transmucosal part of a dental implant, separates the peri-implant bone from the oral cavity. This soft tissue collar is called "peri-implant mucosa". The soft tissue attachment to the implant surface serves as a biological seal that prevents the development of inflammatory peri-implant diseases (i.e. peri-implant mucositis and peri-implantitis) Thus, the soft tissue seal around implants ensures healthy conditions and stable osseointegration and therefore also the long-term survival of an implant. While the soft tissue seal around teeth develops during tooth eruption, the peri-implant mucosa forms after the the surgical wound created to insert the implant. The wound healing phase may occur following the closure of a mucoperiosteal flap around the neck portion of an implant placed in a so-called one-stage procedure or after a second surgical intervention for abutment connections to an already installed dental implant (two-stage procedure).

It seems that the soft tissue adhesion is influenced by the properties (abutment material and micro-topography) of the implant components that are placed in contact with the soft tissues. Abutment material was found to influence bleeding on probing (BoP) at peri-implant soft tissues, as well.

Since wound healing occurs in the presence of a biomaterial (i.e. a foreign body) at a critical region, positive or negative interferences of wound healing events with this biomaterial and adaptation of the soft tissue to this biomaterial have to be taken into consideration. Biocompatibility, soft tissue adhesion, plaque retention, mechanical behavior and esthetics are listed among the criteria of material abutment selection. Titanium remains the most reliable material given its mechanical resistance, biocompatibility, modification of surface increasing cell adhesion and plaque retention. However, in the case of increased esthetics demands, particularly for thin biotype, zirconia and ceramics aluminum abutments give better results with comparable technical and biological outcomes to titanium abutments.

Polyetheretherketone (PEEK) is a strong thermoplastic material produced from polyetheretherketone resin. Because of its high mechanical strength and durability, good electrical characteristics and outstanding resistance to hydrolysis, PEEK has been used extensively in aerospace, automotive, chemical, electronics, petroleum, and food and beverage industries. Recently, a medical-grade PEEK was developed. Medical-grade PEEK has the same physical properties as PEEK; however, PEEK-OPTIMA™ is also biocompatible, has high chemical resistance and resists several different sterilization methods. It is noteworthy to mention that PEEK has an elastic modulus similar to that of the bone preventing marginal bone loss in case of occlusal overload. Due to the aforementioned properties, PEEK has been used as abutment material.

Morphology of the abutment deserves considerations, as well. Some physiological soft-tissue recession can be seen in time around implant restorations when a divergent emergence profile (the most common) is chosen next to the soft tissue. Recently it has been shown how some gingival coronal migration can be seen with the use of tapered emergence profile abutments. In fact, by using these tapered abutments or an implant design with a tapered shape at the neck implant level (transmucosal level), not only soft tissue migration but also hard tissue migration could be achieved over time.

Healing of peri-implant mucosa is characterized by a rapid formation of vascular structures and recruitment of inflammatory cells followed by the maturation of a tissue that eventually establishes a firm barrier of supracrestal connective tissue and long junctional epithelium, which effectively prevents downgrowth of a bacterial biofilm. Angiogenesis as a critical part of wound healing is noticed to peak at 2 weeks with a decline over 10 weeks, while the recruitment of inflammatory cells (B cells and T cells) occur in clusters and decrease from 4 to 8 weeks of healing in connective tissue.

However, little is available on the very early response that might determine the histological organization of peri-implant soft tissues in general and in contact to different macroscopic and microscopically modified materials. Peri-implant soft tissues are part of the gingiva and oral mucosa and implant placement occurs through the creation of an wound. Myofibroblasts represent key players in the physiological reconstruction of connective tissue after injury and in generating the pathological tissue deformations that characterize fibrosis. They constitute a critical cellular source of type I collagen, which is essential during wound healing. Excessive contraction and overproduction of extracellular matrix, mainly collagen, by myofibroblasts can cause tissue fibrosis with formation of hypertrophic scar characterized by reducedtensile strength and disoriented collagen fibres. In full thickness skin wounds, myofibroblast differentiation starts approximately a week after wounding, and contraction peaks at 5-15 days postwounding, but in oral cavity, this step occurs earlier than in skin, given the shorter healing time of these tissues.

Therefore the aim of the present study was to evaluate the myofibroblast component of peri-implant mucosal tissues at different healing abutment materials (titanium gr4, titanium gr 5, zirconium and PEEK) 24 hours after placement.

MATERIALS AND METHODS Ethical aspect This protocol will be evaluated by the Ethical Committee of Sapienza University of Rome after Department approval. Each patient will be provided with a written informed consent.

Study design Biomolecular study of biopsies taken from the peri-implant soft tissue 24 hours after implant and healing abutment placement of four different materials (titanium gr4, titanium gr 5, zirconium and PEEK).

Operators, blindness and allocation Implants and abutments will be placed by a single operator, not involved in other functions during the study. A second operator, not involved in implant or abutment placement, will perform the biopsy. The laboratory operator will be blind of the allocation of biopsies. The type of abutment associated with each implant will be determined in a closed envelope that is going to be opened only when implant is placed. Patients will be informed about the type of implants and abutments used but not about the exact location of each one.

Sample characteristics A total of 10 patients recruited for implant treatment at the Dental clinic of Sapienza University of Rome will participate in the study following the fulfilment of the inclusion and exclusion criteria.

Inclusion criteria:

(I) Age ≥ 18 years (II) Absence of Systemic Diseases / Disorders (III) Smoking ≤ 5 cigarettes per day (IV) Periodontally healthy or treated (V) Full-mouth plaque score (FMPS) ≤ 15% at baseline (VI) Full-mouth bleeding score (FMBS) ≤ 15% at baseline (VII) Presence of edentulous space needing an all on four or all on six treatment with overdenture (VIII) Width of the keratinized gingiva ≥ 2 at the level of the crest

Exclusion criteria: (exclusion of risk / confounding factors):

(I) Pregnancy / lactation (II) Use of systemic antibiotics in the last 3 months (III) Use of systemic antibiotics as prophylaxis for endocarditis (IV) A chronically treated patient (i.e. 2 weeks or longer) with medicines known to affect periodontal tissues (e.g. phenytoin, calcium antagonists, cyclosporine, warfarin and non-steroidal anti-inflammatory drugs) the last month before starting the study (V) Radiotherapy in the neck-head region (VI) HIV, TB, hepatitis or other infectious diseases (VII) Abuse with drugs or alcohol (VIII) Smoked cigarettes> 5 cigarettes per day (IX) Untreated periodontitis (X) FMPS> 15% at baseline (XI) FMBS> 15% at baseline (XII) Implants with peri-implant history (XIII) Width of keratinized tissue over crest <2 mm (XIV) Need for bone reconstruction around implants to be inserted

Clinical treatment

The protocol will follow Tomasi et al 2014 with the modification of a baseline sample taken when incising for the preparation of the flap. Briefly, following local anesthesia, flap elevation and implant placement (Sweden and Martina SpA, Padova, Italy), a specially designed abutment of four different materials (tigran gr4, tigran gr 5, zirconium and PEEK) will be connected to each implant following a double -blinded allocation and flaps will be sutured. Patients will rinse with chlorhexidine for 1 weeks until suture removal. After 24 hours from implant placement, a custum-made cutting device will be used to retrieve a circumferential biopsy of the peri-implant soft tissue. A guide pin will be connected to the abutment and a circular punch with a cutting edge will be forced apically around the abutment dissected a 1.5 mm thick collar of peri-implant soft tissue and removing it together with the abutment and the cutting device. The whole system will be placed in 4% formalin and transferred to a 70% ethanol solution after 48 h.

Cito- histological analysis

Cell Immunofluorescent staining and confocal microscopy. Once harvested with a punch around the implant neck, cells are obtained using the explant method. The 2 mm samples are first minced and then placed in a culture flask and incubated in complete media in 5% CO2 at 37°C. Alternatively, samples are placed in high glucose DMEM supplemented with 15 % FBS and antibiotics, and stored at 4 C for 24 hrs. Cells are then fixed in 4% PFA in PBS for 30 min at room temperature. To label the molecules of interest, the cells are permeabilized in PBS/10% goat serum/0.3% Triton X-100 (1h, 20°C), followed by primary antibodies (against cytoskeletal/cytoskeleton associated proteins and matrix proteins) in PBS/0.1% BSA/0.3% Triton X-100 (4°C, 20°C), washed, and incubated with secondary antibody, DAPI and/or phalloidin (4°C, 20°C). Confocal fluorescence (Leica SP8) and epifluorescence microscopy (DeltaVision system) are performed using 20x/ 0.50 NA and 40x/ 0.80 NA objectives (Olympus FV1000).

Biopsy tissue microscopy. Tissue samples obtained after surgical removal are fixed in formalin and sectioned with a vibratome (Leica, VT100s) to obtain 200 μm thick slices. For optimized antibody penetration, sequential 24 h-incubation (4°C) are performed for each primary and secondary antibody incubation and washing steps (PBS/2% goat serum/0.1% Triton X-100/0.05% NaN3). Images are acquired using two-photon microscopy with a 20x /NA 0.95 objective (Olympus XLUMPlanFI 206) and excitation at 910/1090/1180 nm.

Statistical analysis

A total of 80 samples will be taken at implant insertion and 24 hours after , each analyzed three times. The results will be expressed as mean and SD values and ANOVA and Mann-Whitney test from appropriate software (STATA version 13.1; StataCorp LP; College Station, TX) used to find the difference among the four abutment materials

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Absence of Systemic Diseases / Disorders
* Smoking ≤ 5 cigarettes per day
* Periodontally healthy or treated
* Full-mouth plaque score (FMPS) ≤ 15% at baseline
* Full-mouth bleeding score (FMBS) ≤ 15% at baseline
* Presence of edentulous space needing an all on four or all on six treatment with overdenture
* Width of the keratinized gingiva ≥ 2 at the level of the crest

Exclusion Criteria:

(I) • Pregnancy / lactation

* Use of systemic antibiotics in the last 3 months
* Use of systemic antibiotics as prophylaxis for endocarditis
* A chronically treated patient (i.e. 2 weeks or longer) with medicines known to affect periodontal tissues (e.g. phenytoin, calcium antagonists, cyclosporine, warfarin and non-steroidal anti-inflammatory drugs) the last month before starting the study
* Radiotherapy in the neck-head region
* HIV, TB, hepatitis or other infectious diseases
* Abuse with drugs or alcohol
* Smoked cigarettes> 5 cigarettes per day
* Untreated periodontitis
* FMPS> 15% at baseline
* FMBS> 15% at baseline
* Implants with peri-implant history
* Width of keratinized tissue over crest <2 mm
* Need for bone reconstruction around implants to be inserted

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Early healing of peri-implant soft tissues | 24 hours
  The early healing of soft peri-implant tissues will be interpreted through the activity of myofybroblasts

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pilloni, MD DDS Ms, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Department of Oral and Maxillofacial Sciences. Section of Periodontics.Sapienza, University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindhe J, Wennstrom JL & Berglundh T. The mucosa at teeth and implants. In: Lindhe, J., Lang, N. P. & Karring, T. (eds). Clinical Periodontology and Implant Dentistry, 5th edition, pp. 69-85, 2008.
- [Background] Small PN, Tarnow DP. Gingival recession around implants: a 1-year longitudinal prospective study. Int J Oral Maxillofac Implants. 2000 Jul-Aug;15(4):527-32. PMID 10960986
- [Background] Apse P, Zarb GA, Schmitt A, Lewis DW. The longitudinal effectiveness of osseointegrated dental implants. The Toronto Study: peri-implant mucosal response. Int J Periodontics Restorative Dent. 1991;11(2):94-111. No abstract available. PMID 1718917
- [Background] Rodriguez X, Navajas A, Vela X, Fortuno A, Jimenez J, Nevins M. Arrangement of Peri-implant Connective Tissue Fibers Around Platform-Switching Implants with Conical Abutments and Its Relationship to the Underlying Bone: A Human Histologic Study. Int J Periodontics Restorative Dent. 2016 Jul-Aug;36(4):533-40. doi: 10.11607/prd.2580. PMID 27333011
- [Background] Cocchetto R, Canullo L. The "hybrid abutment": a new design for implant cemented restorations in the esthetic zones. Int J Esthet Dent. 2015 Summer;10(2):186-208. PMID 25874269
- [Background] Braun E, Iacono VJ. Tapered tips to think about. Int J Periodontics Restorative Dent. 2006 Feb;26(1):7. No abstract available. PMID 16515091
- [Background] Urdaneta RA, Leary J, Lubelski W, Emanuel KM, Chuang SK. The effect of implant size 5 x 8 mm on crestal bone levels around single-tooth implants. J Periodontol. 2012 Oct;83(10):1235-44. doi: 10.1902/jop.2012.110299. Epub 2012 Feb 6. PMID 22309172
- [Background] Schwarz F, Mihatovic I, Becker J, Bormann KH, Keeve PL, Friedmann A. Histological evaluation of different abutments in the posterior maxilla and mandible: an experimental study in humans. J Clin Periodontol. 2013 Aug;40(8):807-15. doi: 10.1111/jcpe.12115. Epub 2013 Jun 3. PMID 23725491
- [Background] Waerhaug J. Subgingival plaque and loss of attachment in periodontosis as evaluated on extracted teeth. J Periodontol. 1977 Mar;48(3):125-30. doi: 10.1902/jop.1977.48.3.125. PMID 264960
- [Background] Welander M, Abrahamsson I, Berglundh T. The mucosal barrier at implant abutments of different materials. Clin Oral Implants Res. 2008 Jul;19(7):635-41. doi: 10.1111/j.1600-0501.2008.01543.x. Epub 2008 May 19. PMID 18492075
- [Background] Rompen E, Domken O, Degidi M, Pontes AE, Piattelli A. The effect of material characteristics, of surface topography and of implant components and connections on soft tissue integration: a literature review. Clin Oral Implants Res. 2006 Oct;17 Suppl 2:55-67. doi: 10.1111/j.1600-0501.2006.01367.x. No abstract available. PMID 16968382
- [Background] Sanz-Martin I, Sanz-Sanchez I, Carrillo de Albornoz A, Figuero E, Sanz M. Effects of modified abutment characteristics on peri-implant soft tissue health: A systematic review and meta-analysis. Clin Oral Implants Res. 2018 Jan;29(1):118-129. doi: 10.1111/clr.13097. Epub 2017 Oct 26. PMID 29072346
- [Background] Garcia B, Camacho F, Penarrocha D, Tallarico M, Perez S, Canullo L. Influence of plasma cleaning procedure on the interaction between soft tissue and abutments: a randomized controlled histologic study. Clin Oral Implants Res. 2017 Oct;28(10):1269-1277. doi: 10.1111/clr.12953. Epub 2016 Aug 23. PMID 27552929
- [Background] Tomasi C, Tessarolo F, Caola I, Wennstrom J, Nollo G, Berglundh T. Morphogenesis of peri-implant mucosa revisited: an experimental study in humans. Clin Oral Implants Res. 2014 Sep;25(9):997-1003. doi: 10.1111/clr.12223. Epub 2013 Jun 26. PMID 23799997
- [Background] Linkevicius T, Vaitelis J. The effect of zirconia or titanium as abutment material on soft peri-implant tissues: a systematic review and meta-analysis. Clin Oral Implants Res. 2015 Sep;26 Suppl 11:139-47. doi: 10.1111/clr.12631. Epub 2015 Jun 13. PMID 26073346
- [Background] Sailer I, Philipp A, Zembic A, Pjetursson BE, Hammerle CH, Zwahlen M. A systematic review of the performance of ceramic and metal implant abutments supporting fixed implant reconstructions. Clin Oral Implants Res. 2009 Sep;20 Suppl 4:4-31. doi: 10.1111/j.1600-0501.2009.01787.x. PMID 19663946
- [Background] Neumann EA, Villar CC, Franca FM. Fracture resistance of abutment screws made of titanium, polyetheretherketone, and carbon fiber-reinforced polyetheretherketone. Braz Oral Res. 2014;28:S1806-83242014000100239. doi: 10.1590/1807-3107bor-2014.vol28.0028. Epub 2014 Aug 4. PMID 25098826
- [Background] Steinberg EL, Rath E, Shlaifer A, Chechik O, Maman E, Salai M. Carbon fiber reinforced PEEK Optima--a composite material biomechanical properties and wear/debris characteristics of CF-PEEK composites for orthopedic trauma implants. J Mech Behav Biomed Mater. 2013 Jan;17:221-8. doi: 10.1016/j.jmbbm.2012.09.013. Epub 2012 Oct 11. PMID 23127632